CLINICAL TRIAL: NCT02452008
Title: Overcoming Drug Resistance in Metastatic Castration-resistant Prostate Cancer With Novel Combination of TGF-β Receptor Inhibitor LY2157299 and Enzalutamide: a Randomized Multi-site Phase II Study
Brief Title: Study of TGF-β Receptor Inhibitor Galunisertib (LY2157299) and Enzalutamide in Metastatic Castration-resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Eli Lilly and Company (Industry); National Capital Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J1557; IRB00065746 (Other: JHMIRB)
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: metastatic castration-resistant prostate cancer; enzalutamide; LY2157299; TGF-β receptor inhibitor
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; LY-2157299

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Enzalutamide with LY2157299 (Experimental)
  Interventions: Drug: Enzalutamide; Drug: LY2157299
- Arm 2: Enzalutamide alone (Experimental)
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — 160mg of enzalutamide is administered orally once a day on days 1-28 of each cycle.
  Other Names: XTANDI
Drug: LY2157299 — 150 mg of LY2157299 is administered orally twice a day on days 1-14 of each cycle.
  Other Names: TGF-β receptor inhibitor
  Arms: Arm 1: Enzalutamide with LY2157299

SUMMARY:
The primary objective of this study is to compare the progression free survival (PFS) of patients with metastatic castration-resistant prostate cancer treated with enzalutamide in combination with LY2157299 (Arm 1) versus enzalutamide alone (Arm 2).

ELIGIBILITY:
Inclusion Criteria:

* Have metastatic castration-resistant prostate cancer
* Must have had prior abiraterone treatment
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 2
* Age ≥18 years
* Have measurable disease
* Patients acceptance to have a tumor biopsy of an accessible lesion at baseline and on treatment if the lesion can be biopsied with acceptable clinical risk (as judged by the investigator).
* Ability to take oral medication
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests
* Must use acceptable form of birth control while on study
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Known history or evidence of brain metastases
* Prior chemotherapy for metastatic disease in castration-resistant prostate cancer
* Had surgery within 4 weeks prior to the first dose of study drug
* Had radiation, biological, or other investigational cancer therapy within 2 weeks prior to the first dose of study drug
* Had second-line hormonal therapy within 2 weeks prior to the first dose of study drug
* Systemic steroids within 1 weeks prior to the first dose of study drug
* Had prior enzalutamide, ARN-509, or galeterone therapy
* Have moderate or severe cardiovascular disease
* Have a history of a seizure
* Have uncontrolled intercurrent illness, including but not limited to ongoing or active infection, systematic congestive heart failure, unstable angina pectoris, cardiac arrhythmia or psychiatric condition that would limit compliance with study requirements
* Have a history of any autoimmune disease:inflammatory bowel disease, (including ulcerative colitis and Crohn's Disease), rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythmatosus (SLE) autoimmune vasculitis (e.g., Wegener's Granulomatosis), central nervous system (CNS) or motor neuropathy considered to be of autoimmune origin (e.g., Guillian-Barre Syndrome, Myasthenia Gravis, Multiple Sclerosis)
* Have known history of infection with HIV, hepatitis B, or hepatitis C

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-05-03 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival in patients with metastatic castration-resistant prostate cancer treated with enzalutamide and LY2157299 (Arm 1) versus enzalutamide alone (Arm 2) using RECIST 1.1 criteria. | 4 years

SECONDARY OUTCOMES:
Tumor marker kinetics (PSA) in patients with metastatic castration-resistant prostate cancer treated with enzalutamide and LY2157299 (Arm 1) versus enzalutamide alone (Arm 2). | 4 years
Overall survival (OS) in patients with metastatic castration-resistant prostate cancer treated with enzalutamide and LY2157299 (Arm 1) versus enzalutamide alone (Arm 2). | 4 years
Number of patients experiencing treatment-related toxicities | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Channing Paller, MD, Principal Investigator — Johns Hopkins University
Locations (4):
- United States (4):
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland

REFERENCES:
- [Derived] Rodriguez Y, Unno K, Truica MI, Chalmers ZR, Yoo YA, Vatapalli R, Sagar V, Yu J, Lysy B, Hussain M, Han H, Abdulkadir SA. A Genome-Wide CRISPR Activation Screen Identifies PRRX2 as a Regulator of Enzalutamide Resistance in Prostate Cancer. Cancer Res. 2022 Jun 6;82(11):2110-2123. doi: 10.1158/0008-5472.CAN-21-3565. PMID 35405009